CLINICAL TRIAL: NCT04846244
Title: Real World Effectiveness of Upadacitinib on Early and Sustained Pain Control in Axial Spondylarthritis (UPSTAND)
Brief Title: A Study of the Change in Early and Sustained Pain Control in Axial Spondylarthritis in Adult Participants Receiving Upadacitinib
Acronym: UPSTAND
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-410
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Axial Spondylarthritis (axSpA)
Keywords: Axial Spondylarthritis (axSpA); Upadacitinib; RINVOQ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants Receiving Upadacitinib: Participants receiving Upadacitinib for axial spondyloarthritis (axSpA).

SUMMARY:
Axial spondyloarthritis (axSpA) is an immune-mediated inflammatory disease primarily affecting the axial skeleton. The most frequent axSpA symptom is chronic, often inflammatory back pain (IBP) that might be difficult to distinguish from other causes of chronic back pain (CBP). Many participants report persistent pain, including back pain, which impacts disease activity and quality of life including creating burdens such as sleep disturbance, social isolation, loss of productivity, as well as anxiety and depression. This study will assess the real-world effectiveness of upadacitinib on early and sustained pain control, and the association between pain and clinical/patient-reported outcomes in axSpA participants.

Upadacitinib is being developed for the treatment of axSpA. Approximately 650 adult participants with active-axSpA will be enrolled across approximately 19 countries in Europe, North America, South America, and Asia-Pacific.

Participants will receive oral upadacitinib tablets as prescribed by the physician prior to enrolling in this study in accordance with the terms of the local marketing authorization and professional and reimbursement guidelines with regards to dose, population and indication. Participants will be followed for 12 months.

There may be a higher burden for participants in this study compared to usual standard of care. Participants will attend regular visits per routine clinical practice. The effect of the treatment will be checked by medical assessments, checking for side effects, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Axial Spondylarthritis (axSpA) according to the ASAS criteria.
* Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) score >= 4 at Baseline.
* Total back pain score >= 4 at Baseline.
* Inadequate response to at least two nonsteroidal anti-inflammatory drugs (NSAIDs) over an at least 4-week period in total at maximum recommended or tolerated doses, or participant has an intolerance to contraindication for NSAIDs as defined by the investigator.
* Upadacitinib prescribed in accordance with the applicable approved label and local regulatory and reimbursement policies.

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor.
* Participants demonstrating active symptoms of fibromyalgia as per clinical diagnosis.
* Participation in a clinical trial of an investigational drug, concurrently or within the last 30 days.
* Unwillingness or inability to comply with the study requirements, including completion of patient reported outcome questionnaires.
* Participants who cannot be treated with upadacitinib according to the applicable approved label (e.g., contraindications).
* Vulnerable or protected adult patients with lack of capability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with Radiographic Axial Spondylarthritis (r-axSpA) who have been prescribed upadacitinib in the course of routine practice according to relevant approved licenses.
Sampling Method: Non-Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a Total Spinal Pain Score < 4 and >= 2 Unit (0 - 10) Improvement | Baseline (Week 0) to Week 12
  Total spinal pain consists of the mean of two 0-10 numerical rating scale (NRS) questions: total back pain during the previous week and nocturnal back pain during the previous week.
Percentage of Participants Maintaining Total Spinal Pain < 4 Among Participants Who Achieved Total Spinal Pain < 4 and >= 2 unit (0 - 10) Improvement from Baseline at Week 12 | Week 52
  Total spinal pain score consists of the mean of two 0-10 NRS questions: total back pain during the previous week and nocturnal back pain during the previous week.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (160):
- Argentina (5):
  - Hospital Italiano La Plata /ID# 230779, La Plata, Buenos Aires
  - CER Instituto Medico /ID# 230782, Quilmes, Buenos Aires
  - Instituto CAICI S.R.L /ID# 230781, Rosario, Santa Fe Province
  - Duplicate_CIMER /ID# 230780, San Miguel de Tucumán, Tucumán Province
  - Clinica Regional del Sud /ID# 248866, Río Cuarto
- Australia (8):
  - Paratus Clinical Research Woden /ID# 231460, Phillip, Australian Capital Territory
  - Genesis Research Services /ID# 231593, Broadmeadow, New South Wales
  - Campbelltown Hospital /ID# 231462, Campbelltown, New South Wales
  - Royal Prince Alfred Hospital /ID# 232417, Camperdown, New South Wales
  - BJC Health /ID# 230066, Paramatta, New South Wales
  - Barwon Rheumatology Services /ID# 230068, Geelong, Victoria
  - Peninsula Rheumatology /ID# 240172, Langwarrin, Victoria
  - Joint West Rheumatology /ID# 231461, Murdoch, Western Australia
- Belgium (10):
  - Université Libre de Bruxelles - Hôpital Erasme /ID# 238961, Anderlecht, Brussels Capital
  - Rhumaconsult SPRL /ID# 231439, Charleroi, Hainaut
  - CHU de Liège /ID# 231440, Liège, Liege
  - AZ-Delta /ID# 238966, Roeselare, West-Vlaanderen
  - Onze Lieve Vrouw Hospital /ID# 238963, Aalst
  - AZ Sint-Jan Brugge /ID# 238964, Bruges
  - CHU Brugmann /ID# 238962, Brussels
  - Reumacentrum /ID# 231437, Genk
  - ReumaClinic /ID# 231438, Genk
  - AZ Damiaan /ID# 231441, Ostend
- Bulgaria (5):
  - Prof. Anastas Batalov AIPSMP-VBR EOOD /ID# 249788, Plovdiv
  - Medical center Unimed /ID# 249618, Plovdiv
  - "Ambulatory for individual practice of specialized medical help for internal dis /ID# 249791, Sofia
  - ASIMP Rheumatology Centre "St. Irina" EOOD /ID# 249789, Sofia
  - AIPSMPR -d-r Gerganov /ID# 249749, Varna
- Canada (15):
  - Artus Health Center /ID# 241966, Vancouver, British Columbia
  - Manitoba Clinic /ID# 246217, Winnipeg, Manitoba
  - CIADS Research Co Ltd /ID# 247520, Winnipeg, Manitoba
  - Dr. Juris Lazovskis Inc. /ID# 246574, Sydney, Nova Scotia
  - Dr. Chrisostomos Kouroukis & Dr. Pauline Boulos MPC /ID# 246213, Dundas, Ontario
  - Arthur Karasik Medicine Professional Corporation /ID# 241932, Etobicoke, Ontario
  - Lau Bacchus Professional Medicine Corp /ID# 242591, Hamilton, Ontario
  - Credit Valley Rheumatology /ID# 241948, Mississauga, Ontario
  - The Waterside Clinic /ID# 248678, Orillia, Ontario
  - Dr. Sabeen Anwar Medicine Professional Corporation /ID# 241933, Windsor, Ontario
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 249765, Montreal, Quebec
  - Applied Medical Informatics Research Inc. (AMIR) /ID# 246284, Montreal, Quebec
  - Groupe de Recherche en Maladies Osseuses Inc /ID# 241111, Sainte-Foy, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 247572, Sherbrooke, Quebec
  - Dr Naik-Medical Professional Corporation-Alliance Health /ID# 246516, Saskatoon, Saskatchewan
- France (32):
  - CHU de Besancon - Jean Minjoz /ID# 230528, Besançon, Doubs
  - CHU de Besancon - Jean Minjoz /ID# 242499, Besançon, Doubs
  - Cabinet de rhumatologie /ID# 229091, Mennecy, Essonne
  - CHU Limoges - Dupuytren 1 /ID# 229094, Limoges, Franche-Comte
  - CHU Bordeaux - Hopital Pellegrin /ID# 230548, Bordeaux, Gironde
  - CHU Toulouse - Hopital Purpan /ID# 228818, Toulouse, Haute-Garonne
  - CHU Montpellier - Hôpital Saint Eloi /ID# 228829, Montpellier, Herault
  - CHU Montpellier - Hôpital Saint Eloi /ID# 240980, Montpellier, Herault
  - Polyclinique Courlancy /ID# 229093, Reims, Marne
  - Hopitaux Universitaires Paris Centre-Hopital Cochin /ID# 244006, Paris, Paris
  - CHU de SAINT ETIENNE - Hopital Nord /ID# 228836, Saint Priest EN Jarez, Pays de la Loire Region
  - CHU Nice -Hopital Pasteur /ID# 229088, Nice, Provence-Alpes-Côte d'Azur Region
  - Infirmerie Protestante /ID# 228794, Caluire-et-Cuire, Rhone
  - HCL - Hopital Lyon Sud /ID# 228819, Pierre-Bénite, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 228821, Amiens, Somme
  - CH du Pays d'AIX /ID# 229095, Aix-en-Provence
  - Centre Hospitalier d'Arras /ID# 228833, Arras
  - CHU Clermont Ferrand - Hopital Gabriel Montpied /ID# 229092, Clermont-Ferrand
  - C. H. Sud Francilien /ID# 228826, Corbeil-Essonnes
  - CHD Vendée- La Roche-sur-Yon - Les Oudairies /ID# 230947, La Roche-sur-Yon
  - CHU Grenoble - Hopital Michallon /ID# 228792, La Tronche
  - CHU Lille - Hôpital Roger Salengro /ID# 228820, Lille
  - Clinique de la Sauvegarde /ID# 229087, Lyon
  - Centre Hospitalier Régional d'Orléans - Hôpital de la Source /ID# 234258, Orléans
  - AP-HP - Hopital Saint-Antoine /ID# 228795, Paris
  - Hopital Pitie Salpetriere /ID# 243309, Paris
  - Centre de Soins Osteoarticulaires Ambulatoires /ID# 244737, Paris
  - AP-HP - Hopital Bichat - Claude-Bernard /ID# 228837, Paris
  - GH Diaconesses Croix Saint-Simon /ID# 238548, Paris
  - CHU de Rennes - Hospital Sud /ID# 228842, Rennes
  - Hôpital Charles-Nicolle /ID# 229096, Rouen
  - CH Saint Nazaire /ID# 233186, Saint-Nazaire
- Greece (14):
  - General Hospital of Athens Ippokratio /ID# 241133, Athens, Attica
  - General Hospital of Athens Laiko /ID# 241128, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 241124, Heraklion, Crete
  - 424 General MILITARY Hospital /ID# 241127, Efkarpia (Thessalonikis), Thessaloniki
  - Vougiouklakeio S.A. /ID# 246476, Aigáleo
  - Naval Hospital of Athens /ID# 241129, Athens
  - KAT Atttica General Hospital /ID# 243063, Athens
  - Duplicate_General Hospital of Thessaloniki Agios Pavlos /ID# 243823, Kalamaria
  - Iaso /ID# 245137, Marousi
  - Olympion General Clinic SA /ID# 251794, Pátrai
  - University General Hospital of Patras /ID# 243795, RION Patras Achaia
  - Euromedica Blue Cross Gen Clin /ID# 244945, Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 243796, Thessaloniki
  - Euromedica General Clinic /ID# 241126, Thessaloniki
- Hungary (5):
  - Debreceni Egyetem Klinikai Kozpont /ID# 239936, Debrecen, Hajdú-Bihar
  - Magyar Honvedseg Egeszsegugyi Kozpont /ID# 239939, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz /ID# 239937, Debrecen
  - Hevizgyogyfurdo es Szent Andras Reumakorhaz /ID# 239940, Hévíz
  - Bács-Kiskun Megyei Kórház Szegedi Tudományegyetem AOK Oktató Kórháza /ID# 239938, Kecskemét
- Israel (8):
  - Meir Medical Center /ID# 241868, Kfar Saba, Central District
  - Hillel Yaffe Medical Center /ID# 241869, Hadera, H_efa
  - Bnai Zion Medical Center /ID# 241866, Haifa, H_efa
  - The Lady Davis Carmel Medical Center /ID# 241867, Haifa, H_efa
  - Galilee Medical Center /ID# 241870, Nahariya, Northern District
  - The Baruch Padeh Medical Center Poriya /ID# 249797, Tiberias, Northern District
  - The Chaim Sheba Medical Center /ID# 241305, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 241864, Tel Aviv, Tel Aviv
- Kuwait (5):
  - Adan Hospital /ID# 229679, ADAN
  - Jahra Hospital /ID# 229671, Al Jahra
  - Mubarak Hospital /ID# 250478, Hawalli
  - Mubarak Hospital /ID# 251777, Hawalli
  - Farwaniya Hospital /ID# 231445, Kuwait City
- Mexico (2):
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 238815, Guadalajara, Jalisco
  - Private Office Dr. Orozco /ID# 255210, Guadalajara, Jalisco
- Poland (4):
  - Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im. Wiktora Degi /ID# 243225, Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji /ID# 243232, Warsaw, Masovian Voivodeship
  - Ma?opolskie Badania Kliniczne Sp. z o.o. /ID# 255509, Krakow
  - Jerzy ?wierkot Indywidualna Specjalistyczna Praktyka Lekarska /ID# 244289, Oława
- Russia (19):
  - ChUZ Clinical Hospital RZD-Medicine /ID# 233185, Ulan-Ude, Buryatiya, Respublika
  - Chelyabinsk Regional Clinical Hospital /ID# 244741, Chelyabinsk, Chelyabinsk Oblast
  - Regional Clinical Hospital of Kaliningrad region /ID# 238475, Kaliningrad, Kaliningrad Oblast
  - LLC MC RevmaMed /ID# 238478, Syktyvkar, Komi
  - GBUZ RM Mordovia Republican Central Clinical Hospital /ID# 244738, Saransk, Mordoviya, Respublika
  - Research Institute of Rheumatology named after V.A. Nasonova /ID# 238479, Moscow, Moscow
  - Moscow Regional Research and Clinical Institute n.a. Vladimirskiy (MONIKI) /ID# 232510, Moscow, Moscow Oblast
  - Samara Regional Clinical Hospital n.a. V. D. Seredavin /ID# 231169, Samara, Samara Oblast
  - Nort-Western State Medical University n.a. Mechnikov /ID# 231172, Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital #52 /ID# 238477, Moscow
  - Orenburg State Medical University /ID# 233183, Orenburg
  - Republican hospital named after V.A. Baranov /ID# 231173, Petrozavodsk
  - Clinical Rheumatologic Hospital No 25 /ID# 231171, Saint Petersburg
  - Military Medical Academy n.a. Kirov /ID# 242363, Saint Petersburg
  - Clinic of Samara State Medical University /ID# 241166, Samara
  - Budgetary Institution of the Khanty-Mansiysk Autonomous Okrug-Yugra Surgut Dist /ID# 242369, Surgut
  - Nebbiolo Clinical Research Center /ID# 231167, Tomsk
  - Ulyanovsk Regional Clinical Hospital /ID# 238334, Ulyanovsk
  - Yaroslavl State Medicat University /ID# 231168, Yaroslavl
- Spain (23):
  - Complejo Hospitalario Universitario de Santiago /ID# 249025, Santiago de Compostela, A Coruna
  - Hospital de Mérida /ID# 249037, Mérida, Badajoz
  - Hospital Universitario Germans Trias i Pujol /ID# 249030, Badalona, Barcelona
  - Hospital Universitario Mutua Terrassa /ID# 249031, Terrassa, Barcelona
  - Hospital San Pedro /ID# 249028, Logroño, La Rioja
  - Hospital Universitario Son Llàtzer /ID# 249032, Palma de Mallorca, Las Palmas
  - Hospital Infanta Sofia /ID# 249034, San Sebastián de los Reyes, Madrid
  - Hospital Clinico Universitario Virgen de la Arrixaca /ID# 249042, El Palmar, Murcia
  - Hospital Universitario Canarias /ID# 249043, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Universitario Torrecardenas /ID# 252804, Almería
  - Complejos Hospitalario Universitario de Badajoz /ID# 249036, Badajoz
  - Hospital Campus de la Salud /ID# 252805, Granada
  - Hospital Juan Ramon Jimenez /ID# 249040, Huelva
  - Hospital Universitario de Jaen /ID# 249041, Jaén
  - Hospital Universitario Lucus Augusti /ID# 255820, Lugo
  - Hospital Universitario Ramon y Cajal /ID# 249035, Madrid
  - Hospital Universitario 12 de Octubre /ID# 249033, Madrid
  - Hospital Río Carrión /ID# 249027, Palencia
  - Hospital Universitario Nuestra Señora de Candelaria /ID# 249044, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Macarena /ID# 249039, Seville
  - Hospital Universitario Virgen del Rocio /ID# 249038, Seville
  - Hospital Clinico Universitario de Valladolid /ID# 252001, Valladolid
  - Hospital Virgen de la Concha /ID# 249026, Zamora
- Switzerland (3):
  - Kantonsspital St. Gallen /ID# 230696, Sankt Gallen, Canton of St. Gallen
  - Studio Zanisi /ID# 255681, Locarno, Canton Ticino
  - Rheumatologisches Versorgungszentrum Weinfelden /ID# 239435, Weinfelden, Thurgau
- United Arab Emirates (2):
  - Cleveland Clinic Abu Dhabi /ID# 256292, Abu Dhabi
  - AlAin Hospital /ID# 233803, Dubai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P20-410